CLINICAL TRIAL: NCT02118883
Title: Randomized, Double-blind, Parallel Arm Study of the Effect of Essentia Water, an Electrolyzed High-pH Bottled Water, on Serial Blood Viscosity and Other Hydration Biomarkers in Healthy Subjects
Brief Title: Dehydration, Rehydration, and Blood Viscosity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Essentia Water, LLC (Industry)
Collaborators: Health Onvector Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: ESSHOV102
Record Dates: First submitted 2014-04-16; First posted 2014-04-21 (Estimated); Last update posted 2014-07-16 (Estimated); Status verified 2014-07

CONDITIONS: Dehydration
Keywords: exercise; hydration; dehydration; rehydration; alkaline water; blood viscosity; plasma osmolality; bioimpedance
MeSH Terms: conditions — Dehydration; Motor Activity | interventions — Drinking Water

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Essentia Water (Other): Essentia Water, electrolyzed high-pH water
  Interventions: Other: Essentia Water
- Bottled Water (Other): Purified bottle water
  Interventions: Other: Bottled water

INTERVENTIONS:
Other: Essentia Water
  Other Names: Electrolyzed high-pH water
  Arms: Essentia Water
Other: Bottled water
  Other Names: Purified bottled water
  Arms: Bottled Water

SUMMARY:
The purpose of this study is to examine and compare the rehydration effect of Essentia Water, an electrolyzed high-pH bottled water, with industry-standard bottled water purified by reverse osmosis with minerals added, on (1) whole blood viscosity, (2) plasma osmolality, (3) bioelectrical impedance analysis, and (4) body mass change, using serial measurements in apparently healthy adults following exercise-induced dehydration in a controlled environment.

ELIGIBILITY:
Inclusion Criteria:

* Free from any medication for at least 1 week prior to the study

Exclusion Criteria:

* Any chronic condition requiring regular treatment or medical follow-up
* Bleeding disorder or susceptible to prolonged or uncontrolled bleeding
* Active infection
* Current smoker
* Subject has a BMI equal or greater than 30
* Use of oral contraceptives in the previous 3 months
* Subject is pregnant or breast-feeding
* Currently menstruating

Ages: 25 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2014-04; Primary Completion 2014-06 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Change in whole blood viscosity from dehydrated state | 120 min following rehydration
  Blood viscosity measured using a scanning capillary viscometer

SECONDARY OUTCOMES:
Change in whole blood viscosity from dehydrated state | 15, 30, 60, and 90 min following rehydration
  Blood viscosity measured using scanning capillary viscometer
Change in plasma osmolality from dehydrated state | 15, 30, 60, 90, and 120 min following rehydration
  Plasma osmolality measured using freezing point osmometer
Change in bioelectrical impedance | 45, 75, and 120 min following rehydration
  Impedance is measured to provide an estimation of body composition using a bioelectrical impedance analyzer (RJL Quantum IV).
Body mass change | 45, 75, and 120 min following rehydration

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Fridman, PhD, Principal Investigator — A.J. Drexel Plasma Institute
Locations (1):
- Health Onvector Inc, Camden, New Jersey, United States